CLINICAL TRIAL: NCT06618989
Title: Diagnostic Performance of a Combination of Leukocyte Cell Surface Markers in Predicting the Risk of Severe Bacterial Infection in Febrile Children Under Three Months of Age in the Emergency Department: a Pilot Study. ( CYTOFEB )
Brief Title: Diagnostic Performance of a Combination of Leukocyte Cell Surface Markers in Predicting the Risk of Severe Bacterial Infection in Febrile Children Under Three Months of Age in the Emergency Department: a Pilot Study.
Acronym: CYTOFEB
Status: Recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Pasteur Institute (Unknown); Centre de recherche en épidémiologie et bio statistiques (Unknown); Pitié Salpêtrière Biological Resource Center (Unknown); Centre d'immunologie et des maladies infectieuses (Unknown)
Responsible Party: Sponsor
Other Study IDs: APHP231307
Record Dates: First submitted 2024-09-18; First posted 2024-10-01 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2025-02

CONDITIONS: Children Under 3 Months of Age With Fever
Keywords: fever; diagnostic; severe bacterial infections
MeSH Terms: conditions — Fever; Disease; Bacterial Infections | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood sample
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Blood sampling and follow-up call — An additional 1.5 mL of blood will be collected at the time of the child care in the pediatric emergency department. In addition, a telephone call for patient follow-up (unless still hospitalized) will be done.

SUMMARY:
Fever is a frequent reason for emergency department (ED) visits in infants under 3 months of age. Although viral infections are the most common etiologies, the prevalence of severe bacterial infections (SBI) is high (10%). While in infants with SBI, establishing the diagnosis and initiating rapid intravenous antibiotic therapy is necessary, every effort should be made to avoid it in those at low risk of SBI.

Clinical examination and biomarkers are still sub-optimal for assessing the risk of SBI. As a result, the vast majority of these children receive inpatient intravenous antibiotic therapy.

Flow cytometry is a technique for measuring the expression of biomarkers on the cell surface of leukocytes in response to infection. A French team has identified a combination of some fifteen leukocyte cell surface markers that perform excellently in discriminating between bacterial and viral infections in a population of adults presenting to the emergency department with a suspected infection. However, there are no similar studies in children.

The objective of the study is to assess the diagnostic performance of a combination of biomarkers on the cell surface of leukocytes in discriminating between bacterial and viral infection. Infants less than 3 months of age, visiting the ED for fever will have an extra blood sample in order to measure those biomarkers. The performance of those biomarkers to identify SBI will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Children aged between 7 and 90 days
* Visiting the emergency department with fever (Temperature greater than or equal to 38° measured rectally in the emergency department or reported by parents) OR whose fever is detected during the emergency department visit (Temperature greater than or equal to 38° measured rectally in the emergency department)
* Consent signed by one of the two parents/guardians

Exclusion Criteria:

* Weight less than 2,500 grams
* Chronic illness (heart failure...)
* Known immune deficiency
* Congenital anomaly significantly modifying the probability of bacterial infection (pulmonary malformation, esophageal atresia...)
* Antibiotic therapy in the previous 48 hours
* Clinically evident source of fever: skin infection, joint infection, etc.
* Parents or guardians unable to understand French
* Non-affiliation with a social security scheme (including AME)

Ages: 7 Days to 90 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: All infants aged between 7 and 90 days presenting to emergency departments with fever.
Sampling Method: Non-Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2025-02-24 (Actual); Primary Completion 2026-08-24 (Estimated); Study Completion 2026-09-07 (Estimated)

PRIMARY OUTCOMES:
Diagnostic performance of a combination of leukocyte cell surface markers for identifying IBS in febrile infants under 3 months of age presenting to emergency departments. | At inclusion (D0)
  Diagnostic performance (sensitivity and specificity) of the best performing combination of cell surface markers for identifying BSI in febrile infants under 3 months of age presenting to emergency departments.

CONTACTS AND LOCATIONS:
Overall Officials: Maxime Enault, MD, Principal Investigator — Sorbonne University, hospitalpediatric emergency department, Trousseau hospital
Locations (2):
- France (2):
  - hospitalpediatric emergency department, Trousseau hospital, Paris
  - Sorbonne University, pediatric emergency department, Trousseau hospital, Paris

IPD SHARING:
Plan to Share IPD: Yes
The procedures carried out with the French data privacy authority (CNIL, Commission nationale de l'informatique et des libertés) do not provide for the transmission of the database, nor do the information and consent documents signed by the patients.
  Consultation by the editorial board or interested researchers of individual participant data that underlie the results reported in the article after deidentification may nevertheless be considered, subject to prior determination of the terms and conditions of such consultation and in respect for compliance with the applicable regulations
Supporting Information: Study Protocol, ICF
Time Frame: Beginning 3 months and ending 3 years following article publication. Requests out of these time frame can also be submitted to the sponsor
Access Criteria: Researchers who provide a methodologically sound proposal.